CLINICAL TRIAL: NCT02209545
Title: Buccal Misoprostol Prior to Abdominal Myomectomy for Reduction of Intraoperative Blood Loss: A Randomized Placebo-Controlled Trial
Brief Title: Misoprostol for Reduction of Blood Loss During Fibroid Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was prematurely closed due to low enrollment rates.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Professor in Obstetrics and Gynecology, Reproductive Endo & Infertility, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00091259
Record Dates: First submitted 2014-07-23; First posted 2014-08-06 (Estimated); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Fibroids
Keywords: fibroids, leiomyomata, blood loss, misoprostol
MeSH Terms: conditions — Leiomyoma; Hemorrhage | interventions — Misoprostol; Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Experimental): 25 patients undergoing abdominal myomectomy operation will receive two tablets of misoprostol (400 mcg) buccally one hour before the operation.
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): 25 patients undergoing abdominal myomectomy operation will receive two tablets of Vitamin B6 (100mg) buccally one hour before the operation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — 25 patients undergoing abdominal myomectomy operation will receive two tablets of misoprostol (400 mcg) buccally one hour before the operation.
  Other Names: Cytotec
  Arms: Misoprostol
Drug: Placebo — 25 patients undergoing abdominal myomectomy operation will receive two tablets of Vitamin B6 (100mg) buccally one hour before the operation.
  Other Names: Vitamin B6 (pyridoxine)
  Arms: Placebo

SUMMARY:
The aim of this research work is to assess the impact of a single preoperative dose of buccal misoprostol in reducing blood loss during abdominal fibroid surgery.

DETAILED DESCRIPTION:
This is a trial of women undergoing fibroid surgery at a university-affiliated tertiary care center. Eligible participants will be randomized to receive preoperative 400ucg buccal (under the tongue) misoprostol or placebo on the basis of total fibroid volume, location, parity. Intra-operative blood loss will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for abdominal myomectomy with documented uterine fibroids on pelvic imaging (pelvic ultrasound or MRI) within in last 12 months
* Age ≥ 18 years and ≤ 50 years
* Pre-operative hemoglobin >8 g/dl
* Willing to have buccal administration of misoprostol or a placebo at least one hour pre-procedure.
* Ability to understand and the willingness to sign a written informed consent.
* Admissible medical/surgical history
* Can be previously treated with Depo-Lupron, Depo-Provera, or Oral Contraceptive pills
* Intraoperative use of vasopressin and uterine tourniquet is permissible
* Can have had prior Cesarean delivery

Exclusion Criteria:

* Patients who have had a prior abdominal myomectomy
* Post-menopausal women
* Patients with known bleeding/clotting disorders
* Patients with a history of gynecologic malignancy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to misoprostol
* Any cases converted to abdominal hysterectomy or other additional elective surgical procedures performed at time of abdominal myomectomy will be excluded from data analysis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-10; Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Milad, MD, Principal Investigator — Northwestern University, Northwestern Memorial Hopsital
Locations (1):
- Northwestern University, Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-seven patients enrolled in the study by signing the informed consent form. However, due to the premature closure, not all participants had the opportunity to undergo the intended intervention. Of these, 39 participants successfully completed the intervention, while 8 participants could not undergo the intervention as planned.
Groups:
- Misoprostol: 13 patients undergoing abdominal myomectomy operation will receive two tablets of misoprostol (400 mcg) buccally one hour before the operation.
  Misoprostol: 13 patients undergoing abdominal myomectomy operation will receive two tablets of misoprostol (400 mcg) buccally one hour before the operation.
- Placebo: 26 patients undergoing abdominal myomectomy operation will receive two tablets of Vitamin B6 (100mg) buccally one hour before the operation.
  Placebo: 26 patients undergoing abdominal myomectomy operation will receive two tablets of Vitamin B6 (100mg) buccally one hour before the operation.
Period: Overall Study
Arm/Group | Misoprostol | Placebo
Started | 13 | 26
Completed | 13 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol | Placebo | Total
Number analyzed (Participants) | 13 | 26 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 26 | 39
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 26 | 39
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Estimated Intra-operative Blood Loss
Description: Estimate of blood loss occurring during the surgical procedure as determined by anesthesia staff and documented by anesthesia, nursing and surgical staff as per hospital protocol.
Time Frame: Intra-operative
Population: No data was collected.
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Duration of Procedure
Description: Intra-operative time
Time Frame: Intra-operative
Population: No data was collected.
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Length of Inpatient Hospitalization
Description: Participants will be followed for the duration of their stay, defined as the number of days of post-operative inpatient hospitalization, an expected average of 3 days.
Time Frame: Number of days the patient is hospitalized post-operatively, an expected average of 3 days and a maximum of 90 days post-operatively
Population: No data was collected.
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Post-operative Blood Transfusion
Description: Whether or not a patient receives a post-operative blood transfusion, defined as a transfusion occurring in the immediate post-operative period (during post-operative inpatient hospitalization).
Time Frame: From time of surgery completion through discharge from hospital, an expected average period of 3 days
Population: No data was collected.
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through study completion, an average of 7 years.
Arm/Group | Misoprostol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/26
Other Adverse Events (participants affected / at risk) | 0/13 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT02209545/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT02209545/ICF_001.pdf